CLINICAL TRIAL: NCT01946958
Title: Randomized Control Study of the Impact of Primary Care Triple P on Pediatric Residents and Their Patients
Brief Title: Triple P With Pediatric Residents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: Doris Duke Charitable Foundation (Other)
Responsible Party: Principal Investigator, Fred Rivara, Principal Investigator, Seattle Children's Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: SCH-13683
Record Dates: First submitted 2013-09-06; First posted 2013-09-20 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2013-09

CONDITIONS: Psychosocial Problem; Problematic Behavior in Children; Parenting
Keywords: Triple P

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trained in Primary Care (PC) Triple P (Experimental): This group received standardized training in Primary Care (PC) Triple P.
  Interventions: Behavioral: Training in PC Triple P
- Care as Usal (Experimental): This group provided care as usual. This group was not trained in PC Triple P interventions.
  Interventions: Other: Care As Usual

INTERVENTIONS:
Behavioral: Training in PC Triple P — PC Triple P is a brief parenting intervention combining specific advice from provider with parent rehearsal and self-evaluation.
  Arms: Trained in Primary Care (PC) Triple P
Other: Care As Usual — Pediatric residents not exposed to PC Triple P provide their standard care to parents struggling with parenting issues or child behavior concerns.
  Arms: Care as Usal

SUMMARY:
The objective of this study is to conduct a randomized control trial to evaluate the impact of Triple P on the clinic practice of pediatric residents and on select parent and child outcomes. This study will accomplish that overarching goal through addressing two specific aims.

Aim 1. Triple P's Effect on Pediatric Resident's Practice: test the effect of Triple P training on practice of pediatric residents in addressing and managing psychosocial problems.

Hypothesis 1: At the completion of the trial, residents assigned to the intervention group, compared to residents exposed to the control condition, will have:

1. increased skill levels,
2. increased confidence, and
3. increased satisfaction in dealing with and managing psychosocial issues

Aim 2. Triple P's Effect on Parent and Child Outcomes: test the effect of Triple P interventions on parent's feelings of self efficacy, parent's discipline strategies and on children's externalizing behavior.

Hypothesis 2: At the completion of the intervention, parents and children receiving the intervention, compared to those receiving the control condition, will have:

1. greater reduction in targeted child behavior problems,
2. greater reduction in dysfunctional parenting practices,
3. increased use of appropriate discipline and positive parenting strategies, and
4. greater confidence in parenting ability.

ELIGIBILITY:
Inclusion Criteria for Pediatric Resident:

* Assigned to a participating continuity clinic

Exclusion Criteria for Pediatric Resident:

* Not assigned to a participating continuity clinic

Inclusion Criteria for Parent:

* Parent of an eligible child.
* Speaks English

Exclusion Criteria for Parent:

* A parent of an ineligible child
* Non-English speaking

Inclusion Criteria for Child:

* Treated by a participating resident
* Between 18 months and 12 years old
* Does not have any mental health diagnosis
* Is not receiving medication or therapy from a professional

Exclusion Criteria for Child:

* Not treated by a participating resident
* Age falls outside of eligible range
* Has a mental health diagnosis
* Currently receiving medication or therapy from a professional

Ages: 18 Months to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 155 (Actual)
Dates: Start 2011-07; Primary Completion 2012-06 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change in pediatric resident skills and confidence in conducting parent consultations about child behavior | One year
  Pediatric residents will complete a parent consultation skills and confidence assessment at baseline, pre-training, post-training and follow-up.

SECONDARY OUTCOMES:
Change in family outcomes - parent sense of self efficacy, use of positive discipline and child behavior | One year
  Parents participating in the study will complete an assessment about their discipline strategies, their sense of confidence as a parent and their child's behavior at baseline and follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Frederick P Rivara, MD, MPH, Principal Investigator — Seattle Children's Research Institute, Seattle Children's Hospital, University of Washington